CLINICAL TRIAL: NCT04625777
Title: Acceptability, Feasibility, and Outcomes Testing to Reduce Stress Symptoms Among Clergy
Brief Title: Selah Trial of Stress Interventions for Clergy: Mindfulness Based Stress Reduction, Daily Examen, and Stress Inoculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0238
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Occupational Stress
Keywords: Life Stress; Job Stress; Work-related Stress; Mindfulness; Spiritual
MeSH Terms: conditions — Occupational Stress; Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: The investigators will employ a waitlist preference trial study design. Participants will rank the three interventions and be assigned to their highest-ranking intervention. Participants who rank three interventions equally will be randomly assigned to one of the interventions or the waitlist group. Participants who rank two interventions equally will be randomly assigned to one of their preferred interventions and then randomly assigned to immediate intervention vs waitlist. For the waitlist, participants will be randomly assigned to an intervention with an immediate start of prior to Nov 2020, or to the waitlist control group with a delayed start of Nov 2020 or later. If assigned to the delayed start (a.k.a. waitlist) group, they will be asked for data while waiting (i.e. control group data). The investigators may continue to enroll additional participants following the initial enrollment period and receive their preferred intervention without randomization.
Who Masked: Investigator
Masking Description: The analysis statistician will remain blinded to intervention allocation and waitlist randomized assignment until the analysis plan has been finalized and initial blind reviews have been performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (No Intervention): In this waitlist control condition, participants will not receive any programming intervention. They will know that they have access to stress reduction programming after a certain date. They will also provide survey data at 3 time points and heart rate variability data at 2 time points while waiting. The survey questions will include a wide variety of stress items.
- One of three stress reduction interventions (Experimental): There are three stress reduction interventions: Mindfulness Based Stress Reduction, Daily Examen, and stress inoculation.
  Interventions: Behavioral: Mindfulness Based Stress Reduction; Behavioral: Daily Examen spiritual practice; Behavioral: Stress inoculation combination

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Mindfulness Based Stress Reduction (MBSR) teaches several different kinds of meditation. MBSR is offered as an online course through Duke Integrative Medicine and is based on the national model first developed by Jon Kabat-Zinn at the University of Massachusetts. It includes exercises in awareness of breath, body scans, walking meditation, "choiceless" open awareness, Loving Kindness Meditation, and bringing awareness to the present moment. The MBSR Distance Learning course consists of 8 weekly sessions via video conference and includes meditation instruction, periods of guided practice, and group discussion.
  Arms: One of three stress reduction interventions
Behavioral: Daily Examen spiritual practice — The Daily Examen is a simple but powerful prayer used by Jesuits every day. It takes only 10-15 minutes and can be used to reflect on positive emotions, move past negative emotions, and align one's work with God's work. The Examen directs the person praying to focus on a five-step routine:
  1. Become aware of God's presence;
  2. Give thanks to God for everything in your life;
  3. Review the events of the day guided by the Holy Spirit;
  4. Look at what went well or wrong in the past day; if at fault, ask God for forgiveness; and
  5. Look toward tomorrow - what one thing should you do? Listen to what God is telling you.
  Arms: One of three stress reduction interventions
Behavioral: Stress inoculation combination — This intervention includes a combination of stress inoculation and general stress reduction activities focused on physiology, with exercises that bypass the brain and work directly on the body to mitigate the symptoms of stress. This system is based on Stress Inoculation Training, which uses breathing to prepare people in advance for stressful episodes and recovery skills for following such episodes. The techniques include a variety of breathing, blood flow, and tension control methods, as well as ways to conduct deep tissue massage on oneself to release muscle tension. The awareness aspect involves understanding stress biology and learning to spot the symptoms of stress in oneself and others.
  Arms: One of three stress reduction interventions

SUMMARY:
Certain populations may be particularly susceptible to the adverse effects of chronic stress, particularly chronic work-related stress. One such population is that of clergy doing ministry work. Clergy who are interested in stress reduction will choose one of three interventions: Mindfulness Based Stress Reduction, the Daily Examen, or a set of stress inoculation and breathing exercises called Stress Proofing. The study investigators will examine changes in heart rate variability and self-reported stress symptoms over time among clergy who have participated in one of the three interventions, compared to clergy who have not yet received one of the interventions. The aim of this study is to determine trends in stress outcomes for each of the three interventions. The investigators hypothesize that participation in each intervention will be associated with an improvement in stress outcomes compared to those who have not yet received an intervention.

DETAILED DESCRIPTION:
Certain populations may be particularly susceptible to the adverse effects of chronic stress, particularly chronic work-related stress. One such population is that of clergy doing ministry work. Clergy exhibit high prevalence rates of chronic disease, including diabetes, hypertension, asthma, and joint-related disease, as well as obesity. Further, studies also indicate above-average rates of depression. While no studies directly compare rates of clinical anxiety among clergy versus non-clergy, anxiety rates among clergy are elevated. The high prevalence of physical and mental health issues among clergy may be due in part to stressors from the unique nature of clergy work.

A prominent theory of stress is the job-demand-control-support (JDCS) model, which indicates that stressful jobs are those characterized by high demand, low control, and low support. Clergy perform many demanding roles, including inspiring the congregation, providing one-on-one care for congregants, performing sacraments, educating congregants, overseeing educational programming, and leading social justice activities. The work week typically averages 50 hours or more with the expectation of being on call around-the-clock and the range of skills needed is broad. While certain tasks such as preaching are predictable, clergy have no control over the timing of funerals and congregant crises, and only a variable degree of control over congregant perception of the direction the clergy are taking the congregation. Congregants who are committed to the congregation have strong and often conflicting opinions. In terms of support, clergy experience work-related support to varying degrees; they direct essentially a volunteer workforce and, with the wide range of tasks conducted, they often do not receive the support needed to match the tasks or the emotional challenges faced.

Researchers have developed numerous approaches to manage stress, such as cognitive-behavioral therapy, mindfulness, and relaxation. Not all stress-management interventions are equally effective. Rather, stress-reducing activities are viewed as skills that require regular practice. As such, the most effective interventions are those that individuals are willing and motivated to practice (i.e., patient-preference is an important aspect of evidence-based practice). The current study builds on a pilot study that the investigators conducted with clergy to evaluate the feasibility and acceptability of four potentially stress-reducing interventions while taking participant preference into account. Three of those stress-reducing interventions showed trends of self-reported stress reduction in terms of reduced stress symptoms and/or reactivity to stress. In the current study, the investigators test those three interventions: Mindfulness Based Stress Reduction, the Daily Examen, and a set of stress inoculation and breathing exercises called Stress Proofing.

The study design is a waitlist preferences design. As such, participants choose which of the three interventions they prefer, taking into account the intervention content, format, and scheduling dates. The intervention groups will consist of clergy who sign up for the intervention during the initial recruitment phase and are randomly assigned to start before November 2020. (A secondary per-protocol analysis will include in the intervention groups any clergy who sign up for the intervention after the initial recruitment phase.) The control group will consist of clergy who sign up for the intervention during the initial recruitment phase and are randomly assigned to an intervention start time of November 2020 or later. In addition to random assignment to immediate-start versus delayed-start (waitlist), participants who indicate equal preference for two or more interventions will be randomly assigned to one of their preferred interventions. The investigators' study design allows for testing stress outcomes between those participants who preferred that intervention and those who were waiting for intervention. The design will not allow for comparing outcomes between interventions.

ELIGIBILITY:
Inclusion Criteria:

* Having a current appointment in July 2019 of the North Carolina (NC) Annual Conference or the Western NC Annual Conference of the United Methodist Church (UMC).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Change in self-reported stress symptoms | 12 weeks
  We are using a modified version of the Calgary Symptoms of Stress Inventory and will use continuous mean scores of the overall measure (i.e., all subscales combined). The minimum will be 0 and the maximum 4, with higher scores indicating higher symptoms.
Change in Heart Rate Variability | 12 weeks
  We will collect 48-hour ambulatory heart rate variability (HRV) data using EKG devices.

SECONDARY OUTCOMES:
Change in anxiety symptoms | 12 weeks
  We will use continuous scores (min=0, max=21; higher scores=higher anxiety symptoms) of the Generalized Anxiety Disorder-7 measure.

OTHER OUTCOMES:
Change in perceived stress symptoms | 24 weeks
  We are using a modified version of the Calgary Symptoms of Stress Inventory and will use continuous mean scores of the overall measure (i.e., all subscales combined). The minimum will be 0 and the maximum 4, with higher scores indicating higher symptoms.
Change in anxiety symptoms | 24 weeks
  We will use continuous scores (min=0, max=21; higher scores=higher anxiety symptoms) of the Generalized Anxiety Disorder-7 measure.

CONTACTS AND LOCATIONS:
Overall Officials: Rae Jean Proeschold-Bell, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Proeschold-Bell RJ, Eagle DE, Tice LC, Platt A, Yao J, Larkins JS, Kim ET, Rash JA. The Selah trial: A preference-based partially randomized waitlist control study of three stress management interventions. Transl Behav Med. 2025 Jan 16;15(1):ibae017. doi: 10.1093/tbm/ibae017. PMID 38718169
- [Derived] Proeschold-Bell RJ, Eagle DE, Tice LC, Yao J, Rash JA, Choi JY, Stringfield B, Labrecque SM. The Selah Pilot Study of Spiritual, Mindfulness, and Stress Inoculation Practices on Stress-Related Outcomes Among United Methodist Clergy in the United States. J Relig Health. 2023 Aug;62(4):2686-2710. doi: 10.1007/s10943-023-01848-x. Epub 2023 Jun 26. PMID 37365439
- [Derived] Tice LC, Eagle DE, Rash JA, Larkins JS, Labrecque SM, Platt A, Yao J, Proeschold-Bell RJ. The Selah study protocol of three interventions to manage stress among clergy: a preference-based randomized waitlist control trial. Trials. 2021 Dec 9;22(1):892. doi: 10.1186/s13063-021-05845-x. PMID 34886896
- See also: Study description and recruitment website — https://spiritedlife.org/